CLINICAL TRIAL: NCT00229333
Title: Exploratory Study to Assess the Efficacy of Escitalopram Versus Placebo in the Treatment of Depressive Syndrome in Alzheimer's Disease, Vascular Dementia and Mixed Vascular and Alzheimer's Dementia
Brief Title: Study of Escitalopram Versus Placebo in the Treatment of Depressive Syndrome in Alzheimer's Disease, Vascular Dementia, and Mixed Vascular and Alzheimer's Dementia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-03-3124-AS-CTIL
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Depressive Syndrome
Keywords: Escitalopram; Depression; Dementia; Treatment; Depressive Syndrome in Alzheimer's Disease; Depressive Syndrome in Vascular Dementia; Depressive Syndrome in Mixed Vascular and Alzheimer's Dementia
MeSH Terms: conditions — Depressive Disorder; Depression; Dementia; Alzheimer Disease | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
The goal of the present study is to compare the effectiveness of the active (S)-enantiomer of citalopram, escitalopram with placebo in the treatment of patients with depressive syndrome complicating Alzheimer's dementia (AD), vascular dementia (VD) or mixed dementia (MD), for 8 weeks of double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets criteria for the diagnosis of Alzheimer's dementia, or vascular dementia, or mixed alzheimer's and vascular dementia, according to Diagnostic and Statistical for Mental Disorders, Fourth Edition (DSM-IV) criteria.
* Subject meets the following criteria for depressive syndrome: DSM-IV criteria for major depressive episode; and Cornell Scale of Depression in Dementia is 18 or more.
* The depressive syndrome has been present for at least two weeks preceding study entry (Visit 1).
* The depressive syndrome must be at least moderate in severity at Visit 1 and Visit 2 (cause the subject impairment in functional capacity) and in the opinion of the investigator require pharmacological intervention.
* Score on the Mini Mental State Examination (MMSE) of 10-26 at Visit 1 and at Visit 2.
* Other possible reasons for the subject's depressive symptoms, for example, medications or other medical conditions (such as pain, infection, cancer of the pancreas, etc.), have been excluded as an etiology.

Exclusion Criteria:

General Exclusion Criteria:

* Subjects who need placebo run-in period, and/or their caregivers are unable to comply with Study Period I medication to the extent that drug compliance in the remainder of the study would be compromised as determined by the investigator.
* Investigators, site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Diagnostic Exclusion Criteria:

* Schizophrenia
* Subjects who are judged clinically to be at serious suicidal risk at Visit 1.
* Subjects who have clinically significant psychotic symptoms at Visit 1.
* Subject has a serious neurological condition other than AD, VD or MD including, but not limited to: traumatic (head-brain) dementia, space-occupying lesion, relevant structural abnormalities on brain imaging, etc.
* Subject who underwent CVA for 3 months.
* Subject is doing well on a current antidepressant drug regimen.

Exclusionary Concurrent or Historical Illness:

* Subjects with severe hepatic or renal insufficiency.
* Hypo/hyperthyroidism
* B-12 deficiency

Exclusionary Concomitant or Historical Medications:

* Participation in a clinical trial of another investigational drug within 30 days prior to study entry (Visit 1) and/or any concurrent investigational study.
* Subjects with a history of severe adverse reaction to citalopram or escitalopram.
* Concomitant medication as specified.
* Previous treatment with escitalopram unless, in the opinion of the investigator, the patient's previous treatment was inadequate in dose and/or duration to provide an accurate assessment of the therapy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12

PRIMARY OUTCOMES:
Cornell Scale for Depression in Dementia (CSDD) total score

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI; Cohen-Mansfield et al. 1989)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sverdlik, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel